CLINICAL TRIAL: NCT04164693
Title: Efficacy and Safety of Short-term Postoperative Anticoagulant Therapy to Prevente Thrombosis in Arterovenous Fistula
Acronym: EASOAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yunfeng Xia, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The First ChongQingMU
Record Dates: First submitted 2019-11-09; First posted 2019-11-15 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Thrombosis
Keywords: manitenance hemodialysis; arteriovenous fistula; anticoagulant therapy; fistula function; bleeding risk
MeSH Terms: conditions — Thrombosis; Arteriovenous Fistula | interventions — Heparin, Low-Molecular-Weight; Warfarin

STUDY DESIGN:
Intervention Model Description: The enrolled patients will be randomly assigned to either the anticoagulant group or the control group. Patients in the anticoagulant group will receive a low-dose subcutaneous injection of low molecular weight heparin for the prevention of AVF thrombosis, starting 12-24 hours after the surgery. For patients weighing less than 80kg, enoxaparin sodium 4000IU will be administered once daily, while for those weighing over 80kg, enoxaparin sodium 4000IU will be administered every 12 hours. After discharge, these patients will be switched to oral low-dose warfarin for anticoagulation, with a daily dose of 1.25mg (half tablet) on dialysis days and 2.5mg/day on non-dialysis days. Patients with significantly excessive body weight may be considered for a daily dose of 2.5mg, with a total treatment duration of 4 weeks. Patients in the control group will not receive anticoagulants postoperatively, but both groups will routinely receive antiplatelet therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- anticoagulant group (Experimental): Patients in the anticoagulant group received low-dose subcutaneous injection of low molecular weight heparin for prevention of AVF thrombosis, starting 12-24 hours after surgery. For patients weighing less than 80kg, enoxaparin sodium 4000IU was administered once daily, while for those weighing over 80kg, enoxaparin sodium 4000IU was administered every 12 hours. After discharge, these patients were switched to oral low-dose warfarin for anticoagulation, with a daily dose of 1.25mg (half tablet) on dialysis days, and 2.5mg/day on non-dialysis days. Patients with significantly excessive body weight may be considered for a daily dose of 2.5mg, with a total treatment duration of 4 weeks.
  Interventions: Drug: Low molecular weight heparin
- control group (Other): Patients in the control group did not receive anticoagulants postoperatively, but both groups routinely received antiplatelet therapy.
  Interventions: Other: non anticoagulant therapy group

INTERVENTIONS:
Drug: Low molecular weight heparin — patients began to use low molecular weight heparin or warfarin sodium tablets.
  Other Names: warfarin sodium tablets
  Arms: anticoagulant group
Other: non anticoagulant therapy group — no anticoagulant was used after operation.
  Arms: control group

SUMMARY:
Many guidelines at home and abroad advocate that arteriovenous fistula should be the first choice of permanent vascular access, but it is easy to form thrombus in a short time after arteriovenous fistula molding, resulting in internal fistula stenosis or occlusion. In this study, the investigators plan to screen the patients with arteriovenous fistula in the blood purification center of our hospital. Through the study design of random grouping and open label, the investigators will discuss the use of low molecular weight heparin or warfarin to prevent thrombosis in a short period of time after arteriovenous fistula operation. According to the research results, the investigators will understand efficacy and safety of short-term postoperative anticoagulant therapy to prevente thrombosis in arterovenous fistula.

ELIGIBILITY:
Inclusion Criteria:

* After AVF formation or balloon dilation surgery, there were no significant signs of oozing or bleeding at the surgical incision and operative site observed within 12-24 hours.
* The patient is willing to accept short-term anticoagulant therapy after the surgery, bear related risks, and sign an informed consent form.
* The patient is willing to cooperate with this study, undergo data collection related to the research, and relevant clinical examinations.

Exclusion Criteria.

* Age >80 years;
* Concurrent hematologic diseases that can affect coagulation function;
* Concurrent comorbidities that can affect the patient's bleeding or coagulation functions, such as liver cirrhosis;
* Concurrent active bleeding disorders, such as active gastrointestinal ulcers or active lupus;
* History of major organ bleeding (e.g., intracranial or gastrointestinal) or surgery within the past six months;
* Unwillingness to participate in this study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Blood flow of arteriovenous fistula | up to 12 months
  Blood flow of arteriovenous fistula during hemodialysis from 6 months after operation
arteriovenous fistula dysfunction or occlusion | up to 12 months
  The proportion of arteriovenous fistula dysfunction or occlusion
Active bleeding events | up to 12 months
  such as,bleeding of surgical wound, intracranial, digestive tract and urinary tract, ecchymosis and ecchymosis of skin.
arteriovenous fistula dysfunction or occlusion | up to 12 months
  The time of arteriovenous fistula dysfunction or occlusion
AVF Maturation Failure AVF Maturation Failure AVF Maturation Failure AVF Maturation Failure AVF maturation failure | up to 2 months
  AVF maturation failure two months postoperatively

SECONDARY OUTCOMES:
coagulation index | up to 12 months
  Change of coagulation index
Platelet | up to 12 months
  Changes of platelet indexes
Number of hospitalization | up to 12 months
  Number of hospitalization due to arteriovenous fistula thrombosis.
Death | up to 12 months
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hua Gan, Dr., Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No